CLINICAL TRIAL: NCT06195033
Title: Randomized Controlled Clinical Trial of Internal Fixation of Intertrochanteric Fractures of Femur Guided by Conventional Versus IF-AI Artificial Intelligence Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTH LY IF-AI
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-guided surgical protocol group (Experimental)
  Interventions: Procedure: Surgical protocol guided by artificial intelligence software
- traditional surgical protocol group (No Intervention)

INTERVENTIONS:
Procedure: Surgical protocol guided by artificial intelligence software — At present, the indications for internal fixation of intertrochanteric fractures are not clear. We developed an artificial intelligence software to assist surgeons in determining whether to immobilize lateral and medial posterior wall fractures.
  Arms: AI-guided surgical protocol group

SUMMARY:
Our team has developed an AI software to guide the surgical protocol for femoral intertrochanteric fractures. This is a prospective randomized controlled clinical study that will include patients with femoral intertrochanteric fractures combining medial posterior and lateral wall fractures, and will randomly divide the patients into a traditional surgical protocol group and an AI-guided surgical protocol group. The efficacy and safety indexes such as operation time, blood loss, operation cost, infection rate, hospitalization time, postoperative pain score, fracture healing time, internal fixation failure rate and mortality rate were compared between the two groups to verify the efficacy and safety of AI-guided surgical treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Over 60 years old, male or female.
2. Osteoporosis intertrochanteric fracture, which met the diagnostic criteria of X-ray intertrochanteric fracture, and osteoporosis T-value <2.5.
3. Patients with 1mm resolution CT imaging data.
4. Willing to participate in the project, sign the informed consent, and be able to complete the follow-up work.

Exclusion Criteria:

1. Patients with pathological fractures, old fractures, stress fractures, and periprosthesis fractures;
2. Patients lacking 1mm resolution CT imaging data;
3. Severe malnutrition, heavy smoking, alcoholism and other systemic conditions affect fracture healing;
4. Patients with severe medical diseases that cannot be operated on;
5. Patients participating in other clinical studies.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fracture healing situation 36 weeks after surgery | 36 weeks after surgery
  The results of surgical treatment of the patient were shown by imaging data at 36 weeks after surgery, and the treatment was considered successful without failure of internal fixation.

IPD SHARING:
Plan to Share IPD: No